CLINICAL TRIAL: NCT06187532
Title: Carotid Plaque-Burden Scale and Outcomes. Improvements in Risk Stratification for Future Cardiovascular Disease by Adding to SCORE2. A Real Life Study
Brief Title: Carotid Plaque-Burden Scale and Outcomes. A Real Life Study
Status: Completed | Type: Observational
Sponsor: Fundación para la Formación e Investigación de los Profesionales de la Salud de Extremadura (Other)
Responsible Party: Sponsor
Other Study IDs: 1122023; 11223 (Other: FUNDESALUD)
Record Dates: First submitted 2023-12-14; First posted 2024-01-02 (Actual); Last update posted 2024-02-12 (Actual); Status verified 2023-12

CONDITIONS: Atheroscleroses, Cerebral; Carotid Plaque
Keywords: carotid ultrasound.; Carotid plaque-burden; atheroscleroses events prediction
MeSH Terms: conditions — Intracranial Arteriosclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Carotid ultrasonography has been proposed as a tool for prediction of future cardiovascular disease (CVD). Nevertheless, its role in clinical practice remains controversial.

Methods: The investigators analyse the incidence of CVD and mortality in a cohort of 1004 participants without preexisting CVD according to a simple plaque scale recorded in different segments of the carotid artery assess by ultrasound. A prognostic tool for CV events was development adding Carotid Plaque-Burden (CPB) scale to the Systematic COronary Risk Evaluation (SCORE2) table (CPB- SCORE2 scale).

DETAILED DESCRIPTION:
Based in number of plaques and stenosis a simple plaque scale was recorded in different segments of carotid artery, involving a cohort of 1004 participants with vascular risk factors. Outcomes were recorded during 14 years. A prognostic tool for CV events was development adding simple Carotid Plaque-Burden (CPB) scale to the SCORE2 table (CPB- SCORE2 scale).

ELIGIBILITY:
Inclusion Criteria:

* Any of these vascular risk factors: Total cholesterol >200 mg/dL, hypertension, or diabetes, or receiving medication for them
* No cardiovascular disease: coronary, cerebral o peripheral arterial disease.

Exclusion Criteria:

* Associated conditions: cancer, heart failure, chronic obstructive disease, renal insufficiency, neurodegenerative diseases, rheumatic diseases or chronic infections.
* Neck anatomical barriers to perform ultrasound.
* Enrolled in a clinical trial.
* Attend <70% of regular appointments

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a major vascular risk factor, hypertension, diabetes or hypercholesterolemia, from vascular risk office at the Hospital Universitario San Pedro de Alcántara, Cáceres, Spain
Sampling Method: Non-Probability Sample
Enrollment: 1004 (Actual)
Dates: Start 2000-02-02 (Actual); Primary Completion 2023-04-03 (Actual); Study Completion 2023-12-07 (Actual)

PRIMARY OUTCOMES:
Differences in rates of major adverse cardiovascular events (MACE) | 12 year follow-up
  MACE: number of Major Adverse Cardiovascular Events; myocardial infarction, ictus or amputation or revascularisation of leg due to critical ischaemia
Differences in rates of all-cause death | 12 year follow-up
  All-cause death: number of death from any cause

SECONDARY OUTCOMES:
Diagnostic value of Carotid Plaque-Burden-Systematic COronary Risk EvaluationSystematic COronary Risk Evaluation2 (CPB-SCORE2) table compared to Systematic COronary Risk Evaluation2 (SCORE2) for MACE | 12 year follow-up
  Minimum and maximum values are 1 and 3, were higher scores mean a worse outcome. Sensitivity, Specificity, negative predictive value; positive likelihood ratio; negative likelihood ratio (%). net reclassification index;will be compared between High-Risk vs Low-Intermediate-Risk to PBS-SCORE2 table compared SCORE2.

CONTACTS AND LOCATIONS:
Overall Officials: JUAN SANCHEZ M-TORRERO, PhD, Study Chair — Universidad Extremadura

IPD SHARING:
Plan to Share IPD: No